CLINICAL TRIAL: NCT03154476
Title: Sildenafil for Fontan Associated Liver Disease (SiFALD) Study
Brief Title: Role of Sildenafil for Fontan Associated Liver Disease (SiFALD) Study
Acronym: SiFALD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alexander C. Egbe, Assistant Professor of Medicine and Pediatrics, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 16-008985
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Results first posted 2021-07-28 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-07

CONDITIONS: Cirrhosis; Congenital Heart Disease
MeSH Terms: conditions — Fibrosis; Heart Defects, Congenital | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Randomized Double-blind Placebo-control study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both the treatment arm (sildenafil) and the placebo arm will receive monthly package of similar pills. Equal number of patients will be randomly assigned to each arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sildenafil (Experimental): Subjects randomized to this arm will receive sildenafil 5 mg 3 times per day for the first week, and titrated to 10 mg 3 times per day for the second week, and 20 mg 3 times per day from the third week to the end of the study period, 12 months.
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): Subjects will receive placebo times per day for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — Sildenafil will be initiated at 5 mg 3 times per day for the first week, and titrated to 10 mg 3 times per day for the second week and 20 mg 3 times per day from the third week to the end of the study period, 12 months.
  Other Names: Revatio
  Arms: Sildenafil
Drug: Placebo — Placebo capsules matching study drug
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the medication, sildenafil (also known as Revatio), can slow or stop the progression of liver disease in patients who previously had a Fontan operation.

DETAILED DESCRIPTION:
1. All participants will undergo a baseline liver magnetic resonance elastography. The patients with liver stiffness score >2.5 kiloPascal (KPa) [Normal: ≤2.5 KPa] will be enrolled in the study.
2. In addition to a baseline liver MRE, all participants will undergo cardiac MRI, transthoracic echocardiogram (TTE), FibroSure® (alpha-2 macroglobulin, haptoglobulin, gamma-glutamyltransferase, bilirubin, apolipoprotein A1, and alanine transaminase), and chemistry panel.
3. This will be a double blinded placebo control study design. All participants will be randomized 1:1 to sildenafil or placebo for a total of 12 months therapy.
4. Sildenafil will be initiated at 5 mg 3 times per day for the first week, and titrated to 10 mg 3 times per day for the second week and 20 mg 3 times per day from the 3rd week to the end of the study period. The patients will be required to check their pulse rate and blood pressure daily during the first month of drug therapy. Patient who experience hypotension (blood pressure < 90/50 plus symptoms such as dizziness) during dose titration will be asked to remain on the previous tolerated dose. Patients who cannot tolerate 10 mg 3 times daily will be asked to withdraw from the study and will be asked to continue checking their blood pressure for three days after stopping the medication.
5. After 12 months (+/- 2 weeks) of therapy, all imaging studies (liver MRE, cardiac MRI, TTE) and blood tests (FibroSure® and chemistry panel) will be repeated. A final liver MRE and FibroSure will be performed at 18 months (+/- 2 weeks) for the participants whose 18 months follow-up still falls within the study period.
6. Adverse event and compliance monitoring: During the first month of enrollment (initiation and dose titration), adverse events will be collected by subject report and by weekly telephone interview with dedicated research personnel. For the rest of the study period, adverse events will be collected by subject report and by monthly telephone interview with dedicated research personnel. The research personnel will be responsible for sending out the monthly supply of medications and obtaining a count of the remaining number pills as a measure of compliance. All participants will be provided with a pamphlet containing all the side effects of sildenafil, and contact information of research team for reporting any adverse event of concerns about the study.

ELIGIBILITY:
Inclusion criteria:

* All adult Fontan patients who have no contraindications for magnetic resonance imaging (MRI) will be eligible for the study.

Exclusion criteria:

* Subjects with implantable pacemakers
* Residual cardiac lesions (severe ventricular dysfunction, severe atrioventricular valve regurgitation, Fontan baffle or conduit obstruction)
* Viral hepatitis
* Severe renal dysfunction
* History of sildenafil use in the six months prior to study enrollment
* Ongoing sildenafil therapy
* Patients currently taking nitrates
* Hypotension at baseline (BP <90/50 mmHg)
* Pulmonary veno-occlusive disease
* Hearing/vision impairment
* Pulmonary hypertension due to sickle cell disease
* Women of child-bearing potential with a positive pregnancy test will additionally be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C Egbe, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
The safety of the subject will be monitored throughout the duration of the study. During the first month of enrollment (initiation and dose titration), adverse events will be collected by subject report and by weekly telephone interview with dedicated research personnel. For the rest of the study period, adverse events will be collected by subject report and by monthly telephone interview with dedicated research personnel. All participants will be provided with a pamphlet containing all the side effects of sildenafil, and contact information of research team for reporting any adverse event of concerns about the study.
  The patients will be required to check their pulse rate and blood pressure daily during the first month of drug therapy. Patient who experience hypotension (blood pressure < 90/60 plus symptoms such as dizziness) during dose titration will be asked to remain on the previous tolerated dose

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sildenafil | Placebo
Started | 10 | 10
Completed | 6 | 6
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (6) | 29 (5) | 29 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 7 | 7 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Liver Stiffness as Measured by Magnetic Resonance Elastography (MRE)
Description: Measured using magnetic resonance imaging derived liver stiffness (MRE-LS) reported in kilopascal (kPa).
Time Frame: Baseline, 12 months (52 weeks), 24 months (104 weeks)
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 6 | 6
kPa
  Baseline | 5.69 (0.73) | 5.72 (0.83)
  52 weeks | 5.02 (0.94) | 5.68 (0.74)
  104 weeks | 4.67 (0.86) | 5.74 (0.84)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 24 months on all participants.
Arm/Group | Sildenafil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/76/NCT03154476/Prot_SAP_000.pdf